CLINICAL TRIAL: NCT05058092
Title: The Remedee Solution for Improving the Quality of Life of Fibromyalgia Patients: a Multicenter, Randomized, Controlled Efficacy Trial
Brief Title: Evaluation of the Effectiveness of the Remedee Solution in Fibromyalgia
Acronym: Fibrepik
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Remedee SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Remedee3/Fibrepik
Record Dates: First submitted 2021-09-06; First posted 2021-09-27 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: pain; sleep disturbances; millimeter waves
MeSH Terms: conditions — Fibromyalgia; Pain; Parasomnias

STUDY DESIGN:
Intervention Model Description: Randomization in two groups of type: Immediate Solution vs. Delayed Solution
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Remedee Solution consists of:
  * a wristband designed to deliver millimeter wave
  * a mobile application that allows the patient to follow his treatment sessions
  * a personalized support to improve patient adherence to the technology and to increase compliance and effectiveness of the treatment
  The use of the Remedee Solution start at the randomization day (D0)
  Interventions: Device: Immediate Remedee Solution
- Control (Other): The Remedee Solution consists of:
  * a wristband designed to deliver millimeter wave
  * a mobile application that allows the patient to follow his treatment sessions
  * a personalized support to improve patient adherence to the technology and to increase compliance and effectiveness of the treatment
  The use of the Remedee Solution start at three months (M3) after randomization day
  Interventions: Device: Delayed Remedee Solution

INTERVENTIONS:
Device: Immediate Remedee Solution — * D0 to M3: Remedee Solution + medical care
  * M3 to M6: Remedee Solution without personalized support + medical care
  * M6 to M9: medical care only
  Arms: Intervention
Device: Delayed Remedee Solution — * D0 to M3: medical care only
  * M3 to M6: Remedee Solution + medical care
  * M6 to M9: Remedee Solution without personalized support + medical care
  Arms: Control

SUMMARY:
Fibromyalgia is a chronic and complex condition with symptoms that have a strong impact of patients' quality of life, including musculoskeletal pain, insomnia, fatigue, and stiffness. These symptoms are due to a dysfunction of the central nervous system, namely increased sympathetic and decreased parasympathetic levels of activity, and a deficit in endogenous pain inhibition.

Remedee Labs is developing a unique technology using millimeter waves to stimulate subcutaneous nerve receptors of the wrist, sending a message to the brain, which in turn releases endorphins. These endorphins induce a hypoalgesic effect and activate the parasympathetic nervous system, which reduces pain, stress, and improves sleep.

The Remedee Solution evaluated in this study is a wristband designed to deliver millimeter wave, a mobile application that allows the patient to follow his treatment sessions and a personalized support which aims to improve patient adherence to the technology and to increase compliance and effectiveness of the treatment.

The hypothesis of this study is that regular use of the Remedee Solution for three months improves the quality of life of fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of fibromyalgia according to the American College of Rheumatology criteria (Wolfe et al., 2016),
* FIQ score ≥ 39 (moderate and higher forms) on the day of inclusion (D0),
* with a smartphone that runs on Android 8 and iOS 12 or later,
* agreeing the installation of the Fibrepik app on the smartphone,
* agreeing the collection of the number of steps measured by the smartphone,
* agreeing the installation of the Google Fit app for patients whose smartphone runs on Android (necessary for the collection of the number of steps),
* wrist size compatible with the size M or L of the wristband template,
* affiliated to the social security system or beneficiary of such a system,
* who have signed a consent to participate.

Exclusion Criteria:

* with a characterized depressive episode according to the DSM 5,
* substantial change in treatment in the three months prior to inclusion and in the months to come: change in analgesic level, introduction of a new treatment.
* with a chronic inflammatory pathology (chronic inflammatory rheumatism, rheumatoid arthritis, psoriatic arthritis, spondyloarthritis, lupus,...),
* person in civil proceedings,
* having a dermatological pathology on the wrists, such as oozing dermatosis, hyper sweat or an unhealed lesion,
* with a surgical implant, tattoo or piercing on one of the wrists,
* allergic to metals and/or silicone,
* referred to articles L1121-5 to L1121-8 of the French Public Health Code (CSP): Pregnant, parturient or nursing woman; Person deprived of liberty by judicial or administrative decision; Person subject to a legal protection measure or unable to express his/her consent; Person under psychiatric care
* in a period of exclusion from other interventional research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who significantly improve their fibromyalgia-specific quality of life on the FIQ questionnaire between the inclusion visit at D0 and the 3-month visit (M3). | 3 months
  A decrease in FIQ score ≥ 14% is considered clinically meaningful (Bennett et al., 2009)

SECONDARY OUTCOMES:
Evolution of the quality of sleep between D0 and M3 on the Pittsburg Sleep Quality Index (PSQI) questionnaire. | 3 months
  The score of the PSQI questionnaire is between 0 and 21. The higher score (21) means the worse quality of sleep.
Evolution between D0 and M3 of the average pain score over the week on a Visual Analogic Scale (VAS). | 3 months
  The score of the VAS is beetween 0 and 10. The higher score (10) means the worse pain.
Evolution between D0 and M3 of anxiety and depression on the Hospital and Anxiety Depression scale (HAD). | 3 months
  The HAD scale has two dimensions: anxiety score is between 0 and 21 and depression score is between 0 and 21. The higher score means the worse anxiety or depression.
  To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores:
  * <7 : no symptomatology
  * 8 to 10: doubtful symptomatology
  * >11 : definite symptomatology.
Evolution between D0 and M3 of fatigue between the two groups on the Multidimensional Fatigue Inventory questionnaire (MFI20) | 3 months
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue.
  The score of each dimension is between 4 and 20. Higher score correspond with more acute levels of fatigue.
Evolution of analgesic, antidepressant and sleeping pill intake between D0 and M3 | 3 months
  Patient-reported class, dose and number of analgesic doses, as well as dose and number of antidepressant and sleep medication doses. Both self-prescription and heteroprescription will be counted.
Consumption of care between D0 and M3 | 3 months
  number of:
  * care (procedures, medical consultations, hospitalizations),
  * complementary care (acupuncture, osteopath, naturopath, etc.),
  * psycho-behavioral therapies,
  * complementary treatments (phytotherapy, homeopathy, food supplements).
Evolution between D0 and M3 of the general quality of life on the EQ-5D-5L questionnaire | 3 months
  The EQ-5D-5L is a standardized instrument developped by the Euroquol Group as a measure of health-related quality of life. The EQ-5D-5L contains 5 questions (5Q) with response rated in 5 level (5L) and a visual-analogue-scale between 0 and 100. Responses of the 5 questions results to index.
Evolution between D0 and M3 of physical activity on the Global Physical Activity Questionnaire (GPAC). | 3 months
  Each object has a specific code starting from P1 to P16 and then activity is calculated in MET value. For Work and Recreational domains, Moderate MET value is 4.0 and Vigorous MET value is 8.0 while for Transport domains MET value is 4.0
Evolution of number of steps measured by the subject's smartphone collected from D0 to M3 through the Fibrepik mobile application. | 3 months
Impression of the disease change by the patient on the Patient Global Impression of Change (PGIC) at M3 | 3 months
  The PGIC scale is a 7 point scale depicting a patient's rating of overall improvement.
Impression of the disease change by the caregiver on the Clinician Global Impression of Change (CGIC) scale at M3 | 3 months
  The CGIC scale is a 7 point scale depicting a patient's rating of overall improvement.
Frequency of use of the wristband on the six months of use it | month 6 for Intervention groupe and month 9 for control group
  Analyses of log file of wristband
Usability of the wristband on the modular evaluation of key Components of User Experience (meCUE) questionnaire. | month 6 for Intervention groupe and month 9 for control group
  The questionnaire includes 30 items divided into four independent modules: product perception, emotions, consequence of use and global evaluation.
  For modules 1 to 3, the user indicates his or her level of agreement with statements on a 7-point Likert scale, from "strongly disagree" to "strongly agree.
  The last question of the meCUE (module 4) asks the user to give an overall evaluation of the product on a scale from - 5 (bad) to + 5 (good).
Remedee Solution satisfaction questionnaire (questionnaire created by the sponsor) | month 6 for Intervention groupe and month 9 for control group
  This questionnaire specific to the Remedee Solution includes three parts in order to evaluate the patient's satisfaction with the bracelet, the mobile application and the support. A global score between 0 and 100 is given for each part and qualitative questions allow to better understand this global score
Number, description, classification (serious/non-serious) of adverse effects | 9 months
Outcomes 1 to 12 evaluated at 6 months and at 9 months. | 9 months
  We repeat the measure of outcomes 1 to 12 at 6 and 9 months from the randomization to see the evolution of each of them

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MAINDET, MD, Principal Investigator — University Hospital of Grenoble Alps
Locations (8):
- France (8):
  - University Hospital of Grenoble Alps, Grenoble
  - CHU de Montpellier, Montpellier
  - Cabinet libéral Dr. Lorenzi-Pernot, Mornant
  - Hôpital Lariboisière - Assistance Publique Hôpitaux de Paris, Paris
  - CHU de Rouen, Rouen
  - Hôpital Foch, Suresnes
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Médipôle hôpital mutualiste, Villeurbanne

REFERENCES:
- [Derived] Chipon E, Bosson JL, Minier L, Dumolard A, Vilotitch A, Crouzier D, Maindet C. A drug free solution for improving the quality of life of fibromyalgia patients (Fibrepik): study protocol of a multicenter, randomized, controlled effectiveness trial. Trials. 2022 Sep 5;23(1):740. doi: 10.1186/s13063-022-06693-z. PMID 36064731
- See also: Study protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06693-z